CLINICAL TRIAL: NCT03146728
Title: Finding the Optimal Voluntary Exercise Parameters for Generating a Health Benefit in Those Living With Quadriplegia
Brief Title: Finding the Optimal Voluntary Exercise Parameters for Those Living With Quadriplegia
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Barbara Shay, Associate Professor, University of Manitoba
Other Study IDs: H2011:323; 313540 (Other Grant/Funding Number: CPA-MB)
Record Dates: First submitted 2013-06-14; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Metabolism; Obesity; Spinal Cord Injury
MeSH Terms: conditions — Obesity; Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- tetraplegia, paraplegia: motor complete spinal cord injured individuals with tetraplegia or paraplegia
  Interventions: Other: exercise
- able-bodied: age height and weight matched able bodied
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — energy expenditure will be measured for each of the participants during different conditions, rest, during exercise with the arm crank height high or low. Energy expenditure will also be measured during exercise using different modes (arm ergometer, wheelchair and arm-bike). Results will be compared between rest and exercise and between individuals with SCI and able-bodied.

SUMMARY:
There are over 44,000 persons living with spinal cord injury (SCI) in Canada, who face substantial challenges in maintaining a healthy body composition after injury. As a result, obesity, diabetes and cardiovascular disease are prevalent in this population. Guidelines indicating that twice weekly 20-minute sessions of exercise (plus resistance training) will increase physical fitness in those with SCI have been recently published. However, no SCI-specific guidelines indicating the volume of exercise to reduce the risk of developing obesity-related diseases exist. Longitudinal studies indicate that a weekly exercise-related energy expenditure of 2000 - 2500 Calories is correlated with the least likelihood of cardiovascular disease in the able-bodied population. There is little information regarding energy expenditure (EE) for activities carried out by persons with SCI, with less available for persons with tetraplegia. Once known, this EE data can be used to develop exercise interventions to determine the volume of voluntary exercise required to reduce obesity and risk factors for diabetes and cardiovascular disease in those living with tetraplegia.

DETAILED DESCRIPTION:
In the absence of successful regeneration treatments to recover normal neurological function after spinal cord injury, there has been a needed focus on research aimed at preventing or minimizing the secondary complications of living with a spinal cord injury (SCI). Approximately 44,000 persons live with traumatic spinal cord injury in Canada, half of which have tetraplegia, with 35 new spinal cord injuries (SCI) per million each year. Persons with spinal cord injury SCI are among the most sedentary on the planet, with a much higher incidence of related diseases, such as obesity, glucose intolerance, diabetes and cardiovascular disease than the able-bodied population. At the same time, information needed to minimize the risk of developing these diseases for those living with spinal cord injury is lacking. For example, specific information regarding resting energy requirements, energy expenditure during exercise, and the volume of exercise required to maintain a healthy body composition and prevent the development of sedentary-related disease in this population is scarce.

In order to maintain weight, and not gain excess body fat, energy intake in food Calories needs to match energy use. In addition to understanding energy use in order to maintain weight balance, exercise is also important for muscular and cardiovascular health. Research to date indicates that the resting energy expenditure of persons with SCI is considerably less than able-bodied persons with the same weight or body mass index. A considerable portion of this reduced resting energy expense is due to the reduced muscle mass after SCI. There are mixed research results regarding whether there are additional reductions in resting energy expenditure, after adjusting for fat free mass, in persons with SCI. Training has been shown to be effective in reducing shoulder pain, improving function, improving physical capacity, reducing hyperinsulinemia, and reducing dyslipidemia in persons with chronic paraplegia.

However, it is less clear if voluntary exercise can have the same beneficial effects for those living with tetraplegia, in part because their peak power output is only one-third to one-half that achieved during arm exercise in those with paraplegia. In addition, it may be very difficult for those with tetraplegia to be able to exercise for a sufficient duration to achieve a sufficient training effect to either maintain a healthy body composition or reduce the risk of developing the sedentary diseases common to this population. This study will provide the exercise-related energy expenditure data to address this question.

ELIGIBILITY:
Inclusion Criteria:

* motor complete spinal cord injury
* tetraplegia or paraplegia
* stabile condition

Exclusion Criteria:

* serious overuse injuries of the upper extremities
* known cardiovascular disease
* current pressure ulcers
* morbid obesity
* known thyroid dysfunction
* cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will consist of 7 persons living with tetraplegia in addition to 7 persons living with paraplegia to act as controls for study 1. Participants will have sustained a motor-complete spinal cord injury at least 6 months previous. Able-bodied participants are matched for age, height and weight.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
changes in energy expenditure | At baseline, and every minute for three minutes of steady state exercise
  Study 1 will test if optimizing the height of the arm crank axis during arm cycle ergometry will show a greater mechanical efficiency for those with tetraplegia and lead to a longer duration of sustained rhythmic exercise.
  Study 2 will determine the energy expenditure while performing different modes and intensities of voluntary exercise in those with tetraplegia (wheeling, arm cycle ergometry and hand-cycling).
  Study 3: Will determine if periods of reduced core temperature are present and contribute to the reduced basal and resting energy expenditure in those living with tetraplegia.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Shay, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada